CLINICAL TRIAL: NCT00317603
Title: A Phase I Trial of Vaccination With Autologous, Lethally Irradiated Breast Cancer Cells Engineered by Adenoviral Mediated Gene Transfer to Secrete Granulocyte-Macrophage Colony Stimulating Factor in Metastatic Breast Cancer Patients
Brief Title: Vaccination With Autologous Breast Cancer Cells Engineered to Secrete Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) in Metastatic Breast Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Ana C Garrido-Castro, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-111
Record Dates: First submitted 2006-04-21; First posted 2006-04-25 (Estimated); Results first posted 2021-10-14 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer
Keywords: autologous vaccination; GM-CSF; adenoviral mediated gene transfer; Stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms

ARMS (1):
- Vaccine (Experimental): Vaccinations will be administered on days 1,8,15 and every two weeks thereafter until the supply of vaccine has been exhausted or the patient is removed from study. As indicated in 5.2.5, vaccine cell dosage will be approximately 1x10 7 , 4x10 6 ,
  1x10 6 , or 1x10 5 depending on the final cell yield.
  Interventions: Biological: Autologous, Lethally Irradiated Breast Cancer Cells

INTERVENTIONS:
Biological: Autologous, Lethally Irradiated Breast Cancer Cells — Vaccine will be administered on days 1, 8, 15, 29 and then every 2 weeks until the supply of vaccine runs out

SUMMARY:
The purpose of this trial is to test the safety of a vaccine made from a patient's own breast cancer cells, and determine if this vaccine will delay or stop the growth of the cancer. The vaccine is made by genetically modifying a patient's own tumor cells to secrete granulocyte-macrophage colony-stimulating factor (GM-CSF) to activate the immune response.

DETAILED DESCRIPTION:
After the patient has given their consent to participate in the trial, a series of tests will be performed to determine if the patient is eligible. These tests may take place up to 21 days before the surgery to remove a tumor sample or cancer-containing fluid, which will be used to create the vaccines. The tumor cells or fluid is then brought to a special, certified laboratory where the vaccine is made. Specially trained laboratory technicians then use a method known as adenoviral mediated gene transfer, which adds a new gene to the cancer cells. This gene causes the cells to make GM-CSF, a powerful hormone that stimulates the immune system. The cells are then given radiation so that they will not grow. Participants will start receiving vaccine on day 1, 8, 15, 29, and then every two weeks until the supply of vaccine has run out. The amount of the vaccine depends upon the total amount of cells that are obtained from the breast cancer tumor or fluid. Each time the patient is vaccinated, they will be given injections that will be placed underneath the skin. A different place will be used for each injection. If there are enough cells from the patient's tumor sample, the patient will be given an injection of non-transduced irradiated cells (the gene was not added) . These cells will help to measure how the patient's immune system is reacting to the tumor cells. This is called Delayed-Type Hypersensitivity (DTH). With vaccine #1 and #5, the patient will also receive a DTH injection. Two to three days after the vaccine and DTH injection, skin biopsies will be taken of both sites. At week 10 in the study treatment, or earlier if necessary, the patient will have a chest, abdomen, and pelvic CT scan to determine if the vaccine therapy has had an effect on their disease. A brain MRI will be performed if there were any abnormalities on the first brain MRI or if new symptoms have developed. Patients may participate in this study until one of the following happens: All vaccine created from the tumor has been given to the patient; the patient's disease worsens; the patient experiences an unacceptable and/or harmful side effect; the patient is unable to follow the study plan; or the patient's doctor feels it is no longer in the best interest of the patient to continue.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Stage IV breast cancer
* Prior banked malignant effusion or significant malignant effusion for tumor harvest or surgically-accessible tumor nodule of at least 2cm in greatest diameter by physical exam, magnetic resonance imaging (MRI) or computed tomography (CT) scan
* Must have received at least one prior regimen of chemotherapy for metastatic disease
* Patients with HER2 positive tumors must have received at least one prior trastuzumab-based therapy in the metastatic setting, and may not receive trastuzumab therapy and vaccine treatment concurrently
* Patients may receive concurrent bisphosphonate therapy and/or erythropoetin therapy at any point while on study
* ECOG performance status 0 or 1
* Estimated life expectancy of greater than or equal to 6 months
* 18 years of age or older
* Greater than 4 weeks from immunotherapy, or systemic glucocorticoid therapy
* Adequate recovery from drug-related toxicities from prior systemic therapies
* Adequate recovery from recent surgery and radiation therapy
* Greater than 6 months since bone marrow or peripheral blood stem cell transplant

Exclusion Criteria:

* Urgent need for cytotoxic chemotherapy, radiotherapy, or surgery in the next 60 days
* Uncontrolled active infection or illness
* Psychiatric illness/social situation that would limit study compliance
* Pregnant or nursing mothers
* Evidence of HIV infection
* Previous participation in an adenovirus-based trial
* Concurrent invasive malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2008-05 (Actual); Study Completion 2021-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth Overmoyer, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Anderson KS, Erick TK, Chen M, Daley H, Campbell M, Colson Y, Mihm M, Zakka LR, Hopper M, Barry W, Winer EP, Dranoff G, Overmoyer B. The feasibility of using an autologous GM-CSF-secreting breast cancer vaccine to induce immunity in patients with stage II-III and metastatic breast cancers. Breast Cancer Res Treat. 2022 Jul;194(1):65-78. doi: 10.1007/s10549-022-06562-y. Epub 2022 Apr 28. PMID 35482127

RESULTS

PARTICIPANT FLOW:
Recruitment Details: January 2006 through May 2008
Groups:
- Vaccine: Vaccinations will be administered on days 1,8,15 and every two weeks thereafter until the supply of vaccine has been exhausted or the patient is removed from study. As indicated in 5.2.5, vaccine cell dosage will be approximately 1x10 7 , 4x10 6 ,
  1x10 6 , or 1x10 5 depending on the final cell yield.
  Autologous, Lethally Irradiated Breast Cancer Cells: Vaccine will be administered on days 1, 8, 15, 29 and then every 2 weeks until the supply of vaccine runs out
Period: Overall Study
Arm/Group | Vaccine
Started | 15
Treated | 12
Completed | 12
Not Completed | 3
Not completed — Progressive Disease | 3

BASELINE CHARACTERISTICS:
Population: Analysis Population includes only enrolled and treated participants.
Arm/Group | Vaccine
Number analyzed (Participants) | 12
Age, Continuous [Mean (Full Range); unit: years] | 51.5 [34 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Site of Disease [Count of Participants; unit: Participants]
  Skin / Lymph Nodes | 9
  Pleura | 8
  Bone | 9
  Viscera | 9
  Central Nervous System | 1
  Ascites | 1
  Chest Wall | 1
Median Duration of Stage IV Breast Cancer [Median (Full Range); unit: years] | 3.45 [0.4 to 12]
Hormone Receptor Status [Count of Participants; unit: Participants]
  Positive | 8
  Negative | 4
Human Epidermal Growth Factor Receptor 2 Status [Count of Participants; unit: Participants]
  Positive | 5
  Negative | 7
Median number of prior lines of chemotherapy in the metastatic setting (range) [Median (Full Range); unit: therapies] | 2.5 [1 to 7]

OUTCOME MEASURES:

1. Primary Outcome: Minimum Number of Vaccine Doses Created Using Participant Tumor Sample
Description: Tumor samples were obtained via malignant effusion or a surgically accessible tumor nodule of 2 cm in greatest diameter. Tumor cells were processed to single cell suspension and transduced with adenoviral vector encoding human Granulocyte-macrophage colony-stimulating factor (GM-CSF). Then, the cells washed extensively and irradiated with 10,000 cGy. Over the next 14 days, sterility cultures were tested for endotoxin and mycoplasma contamination. Individual vaccine cell dose and number varied depending on the final cell yield from vaccine production. The minimal dose was 1 x 10^5 cells and the maximal dose was 1 x 10^7 cells.
Time Frame: Vaccine doses created and banked soon after registration, up to 8 days.
Population: Vaccinations prepared for "enrolled for vaccine administration" population.
Measure: Number; unit: doses
Arm/Group | Vaccine
Number analyzed (Participants) | 12
doses | 6

2. Secondary Outcome: Number of Participants With Grade 3 or Higher Adverse Events
Description: Number of participants with grade 3 or higher adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: Up to 58 Months
Population: Analysis population for adverse events is "Treated" population.
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine
Number analyzed (Participants) | 12
Participants
  Grade 3 | 0
  Grade 4 | 0
  Grade 5 | 0

3. Secondary Outcome: Number of Participants With RECIST Criteria Responses
Description: Clinical outcomes as measured by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. For target lesions, complete response (CR) is complete disappearance of all target lesions and partial response (PR) is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. Progressive disease (PD) is at least a 20% increase in sum LD of target lesions (smallest sum LD reference), new lesions, and/or unequivocal progression of existing non-target lesions. Stable disease (SD) is defined as any condition not meeting the above criteria.
Time Frame: Up to 14 Years
Population: Clinical outcomes assessed for the "treated" population.
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine
Number analyzed (Participants) | 12
Participants
  Progressive Disease within 2 months | 8
  Stable Disease with progression at 4 months | 2
  Stable Disease with progression at 13 months | 1
  No Evidence of Disease > 12 years | 1

ADVERSE EVENTS:
Time Frame: 14 Years
Description: Serious AEs (SAE) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. All remaining AEs are classified as Other AEs (OAE) including grade 3 or higher events with treatment-attribution of unlikely and unrelated plus all grade 1 and 2 events. Maximum grade toxicity by type was then calculated within SAE and OAE datasets. No further data is available to specify classification of other beyond the general term.
Arm/Group | Vaccine
All-Cause Mortality (participants affected / at risk) | 12/12
Serious Adverse Events (participants affected / at risk) | 3/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccine (N=12)
Hemoglobin (Blood and lymphatic system disorders) | 1
Alkaline phosphatase (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Syncope (Nervous system disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccine (N=12)
Hemoglobin (Blood and lymphatic system disorders) | 8
Palpitations (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 4
Distention/bloating, abdominal (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 7
Lip, pain (Gastrointestinal disorders) | 8
Fatigue (General disorders) | 10
Fever w/o neutropenia (General disorders) | 4
Rigors/chills (General disorders) | 1
Injection site reaction (General disorders) | 8
Edema head and neck (General disorders) | 1
Edema limb (General disorders) | 8
Chest/thoracic pain NOS (General disorders) | 1
Pain NOS (General disorders) | 1
Infection Gr0-2 neut, sinus (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Leukocytes (Investigations) | 6
Lymphopenia (Investigations) | 1
Neutrophils (Investigations) | 3
Platelets (Investigations) | 2
Alkaline phosphatase (Investigations) | 6
ALT, SGPT (Investigations) | 3
AST, SGOT (Investigations) | 6
Bilirubin (Investigations) | 1
Creatinine (Investigations) | 1
Vital capacity (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 8
Hypercalcemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypernatremia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Lumbar spine-range of motion (Musculoskeletal and connective tissue disorders) | 1
Back, pain (Musculoskeletal and connective tissue disorders) | 3
Bone, pain (Musculoskeletal and connective tissue disorders) | 1
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 1
Joint, pain (Musculoskeletal and connective tissue disorders) | 1
Muscle, pain (Musculoskeletal and connective tissue disorders) | 2
Neck, pain (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 3
Neuropathy-sensory (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 1
Head/headache (Nervous system disorders) | 4
Insomnia (Psychiatric disorders) | 4
Proteinuria (Renal and urinary disorders) | 1
Urinary frequency/urgency (Renal and urinary disorders) | 2
Breast, pain (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3
Throat/pharynx/larynx, pain (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Dry skin (Skin and subcutaneous tissue disorders) | 1
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 6
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes